CLINICAL TRIAL: NCT01497405
Title: Combination Prevention for Vulnerable Women in South Africa
Brief Title: WHC+ (Women's Health CoOp PLUS)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: RTI International (Other)
Collaborators: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1R01DA032061-01 (NIH)
Record Dates: First submitted 2011-12-01; First posted 2011-12-22 (Estimated); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: HIV; Sexual Risk; Sexually Transmitted Diseases; Substance Abuse; Violence; Victimization
Keywords: Gender-based Violence; HIV; Randomized Controlled Trial; Sexually Transmitted Diseases; Substance Abuse Detection; Test, Treat and Retain
MeSH Terms: conditions — Sexually Transmitted Diseases; Substance-Related Disorders | interventions — Coal Tar; Single Person

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Test, Treat, Retain(TTR) only (Active Comparator): Participants in this group will be screened for HIV. HIV positive women will be given post-test counseling and referrals for prompt medical evaluation.
  Interventions: Biological: Test, Treat, Retain(TTR) only
- Test, Treat, Retain(TTR) + Women's Health CoOp (WHC) (Experimental): TTR +WHC: Participants in this group will be screened for HIV. HIV positive women, will be given post-test counseling and referrals for prompt medical evaluation and assessment. Both HIV negative and positive participants in this group will participate in 2 individual behavioral counseling sessions focusing on reducing HIV risk behaviours, alcohol and other drug use, and risk of violent victimization. It also adds case management to increase follow through with referrals and risk reduction plans and activities. This intervention is an adaptation of the evidence-based Women's CoOp(PI: Dr. Wendee M. Wechsberg).
  Interventions: Behavioral: Test, Treat, Retain(TTR) + Women's Health CoOp (WHC)

INTERVENTIONS:
Behavioral: Test, Treat, Retain(TTR) + Women's Health CoOp (WHC) — TTR +WHC: Participants in this group will be screened for HIV. HIV positive women, will be given post-test counseling and referrals for prompt medical evaluation and assessment.Both HIV negative and positive participants in this group will participate in 2 individual behavioral counseling sessions focusing on reducing HIV risk behaviours, alcohol and other drug use, and risk of violent victimization. It also adds case management to increase follow through with referrals and risk reduction plans and activities.This will also include case management sessions. This intervention is an adaptation of the evidence-based Women's CoOp (PI: Dr. Wendee M. Wechsberg).
  Arms: Test, Treat, Retain(TTR) + Women's Health CoOp (WHC)
Biological: Test, Treat, Retain(TTR) only — TTR +only: Participants in this group will be screened for HIV. HIV positive women will be given post-test counseling and referrals for prompt medical evaluation.
  Arms: Test, Treat, Retain(TTR) only

SUMMARY:
This study compares the effects of standard HIV test, treat and retain (TTR) practices with TTR plus a woman-focused enhanced strategy--Women's Health CoOp (WHC+) intervention) targeting hard-to-reach and vulnerable alcohol and other drug (AOD)-using women to determine if the WHC+ intervention is more efficacious than TTR alone in reducing HIV risk behavior. Additionally, the study will determine whether HIV positive women in the WHC+ arm are more likely to follow through with referrals for further medical evaluation and linkages to HIV treatment and other care than women in the TTR arm.

DETAILED DESCRIPTION:
There is growing recognition that no single strategy will be sufficient to eliminate transmission. In light of evidence that neither existing biomedical interventions nor any existing behavioral interventions will be sufficient to control the HIV epidemic in South Africa, the proposed study will combine a biomedical intervention with an evidence-based behavioral intervention (i.e., the Women's Health CoOp) to maximize the efficacy of both strategies. If this combination intervention proves efficacious, there is a high likelihood that it can be widely implemented, be sustainable and have a substantial public health impact by reducing the exceedingly high HIV incidence in South Africa.

The overarching goal of the proposed research is to determine whether this enhanced combination prevention strategy targeting vulnerable AOD-using women is more efficacious than current standard practices. The specific aims of the proposed study are:

Aim 1: To expand the WHC outreach strategies to reach more alcohol and other drug (AOD) - using vulnerable women in Pretoria, South Africa.

Aim 2: To test whether adding WHC to standard Treat, Test, and Retain (TTR) practices results in more HIV-positive AOD-using women getting medical evaluations (e.g., cluster of differentiation 4 (CD4), viral load), starting treatment, staying in treatment and in greater reductions in risk behaviors (e.g., AOD use, condom use, victimization) among all women-positive or negative.

The study uses a geographical cluster randomized design. Hotspots (i.e. places where sex workers and drug using women congregate) in the city of Pretoria and the surrounding areas were mapped using geographic information system (GIS) software. Fourteen hotspots were identified and geocoded. The entire area was divided into 14 zones, each of which included a hotspot. Seven matched pairs of zones were created based on socio-economic conditions and estimates of the numbers of sex workers and drug-using women residing in them. Zones within pairs were randomized to the TTR arm or the WHC+ arm. Participants are recruited by outreach workers and their intervention condition is based on the zone from which they were recruited. At study enrollment/baseline, eligible participants complete a questionnaire and baseline HIV, drug and pregnancy testing. Follow-up data collection will be conducted at 6-months and 12-months post-baseline.

ELIGIBILITY:
Inclusion Criteria:

1. Female
2. Black/African
3. 15 years or older (if under 18, must be able to sign assent)
4. Use at least one of the following drugs: alcohol, marijuana (dagga), methamphetamine (tik), Mandrax (methaqualone), cocaine (crack and/or powder), heroin (Thai White), inhalants (glue and benzene) methylenedioxymethamphetamine (MDMA -ecstasy), lysergic acid diethylamide (LSD), or Kat/cat, Nyaope (a mixture of marijuana and heroin) - weekly in the past 90 days
5. Have had unprotected vaginal sex with a male partner in the last six months
6. Able to speak English, Sesotho, Tswana, or Zulu
7. Consent to HIV rapid testing and drug testing
8. Provide written verbal and assent/consent to participate
9. Able to provide verifiable locator information for the Tshwane area and plan to stay there in the next 12 months

Exclusion Criteria:

1. Males
2. Individuals who do not self-identify as Black/African

Ages: 15 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 641 (Actual)
Dates: Start 2012-05; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Unprotected intercourse among women | 6 months
  Percentages of condom use at last sex
Unprotected intercourse among women | 12 months
  Percentages of condom use at last sex

SECONDARY OUTCOMES:
Medical evaluation initiation amongst HIV-positive | 6 months
  Percentages of HIV-positive women receiving medical evaluations.
Medical evaluation initiation amongst HIV-positive | 12 months
  Percentages of HIV-positive women receiving medical evaluations.
Treatment initiation and retention amongst HIV-positive women | 6 months
  Percentages of HIV-positive women starting and staying in treatment
Treatment initiation and retention amongst HIV-positive women | 12 months
  Percentages of HIV-positive women starting and staying in treatment
HIV viral load among HIV-positive women who meet criteria for antiretroviral treatment (ART) and who produce medical records with HIV viral loads | 6 months
  HIV viral load from medical record
HIV viral load among HIV-positive women who meet criteria for antiretroviral treatment (ART) and who produce medical records with HIV viral loads | 12 months
  HIV viral load from medical record
Alcohol use | 6 months post intervention
  Frequency of alcohol use in previous 30 days measured by Revised Risk Behavior Assessment (RRBA) and breath test
Alcohol use | 12 months post intervention
  Frequency of alcohol use in previous 30 days measured by Revised Risk Behavior Assessment (RRBA) and breath test
Victimization | 6 months post intervention
  Percentages of women who report being beaten, attacked with a weapon, or forced to have sex in the previous 90 days
Victimization | 12 months post intervention
  Percentages of women who report being beaten, attacked with a weapon, or forced to have sex in the previous 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Felicia Browne, ScD, Principal Investigator — RTI International
Locations (2):
- RTI International - Headquarters, Research Triangle Park, North Carolina, United States
- Wesley Community Centre, Pretoria, South Africa

REFERENCES:
- [Background] Wechsberg WM, Deren S, Myers B, Kirtadze I, Zule WA, Howard B, El-Bassel N. Gender-Specific HIV Prevention Interventions for Women Who Use Alcohol and Other Drugs: The Evolution of the Science and Future Directions. J Acquir Immune Defic Syndr. 2015 Jun 1;69 Suppl 2(0 1):S128-39. doi: 10.1097/QAI.0000000000000627. PMID 25978479
- [Derived] Wechsberg WM, Peasant C, Kline T, Zule WA, Ndirangu J, Browne FA, Gabel C, van der Horst C. HIV Prevention Among Women Who Use Substances And Report Sex Work: Risk Groups Identified Among South African Women. AIDS Behav. 2017 Nov;21(Suppl 2):155-166. doi: 10.1007/s10461-017-1889-0. PMID 28887751
- [Derived] Wechsberg WM, van der Horst C, Ndirangu J, Doherty IA, Kline T, Browne FA, Belus JM, Nance R, Zule WA. Seek, test, treat: substance-using women in the HIV treatment cascade in South Africa. Addict Sci Clin Pract. 2017 Apr 26;12(1):12. doi: 10.1186/s13722-017-0077-x. PMID 28441975
- [Derived] Wechsberg WM, Zule WA, Ndirangu J, Kline TL, Rodman NF, Doherty IA, Novak SP, van der Horst CM. The biobehavioral Women's Health CoOp in Pretoria, South Africa: study protocol for a cluster-randomized design. BMC Public Health. 2014 Oct 15;14:1074. doi: 10.1186/1471-2458-14-1074. PMID 25318563